CLINICAL TRIAL: NCT04412993
Title: Evaluation of ABO Isoagglutinins Level in Blood Group O Donors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RH Ahmed, RH Ahmed, Assiut University
Other Study IDs: ABO isoagglutinin
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Isoagglutinins Level
Keywords: urgent blood transfusion , group O

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: withdraw blood samples — withdraw blood sample from gorup O donors

SUMMARY:
Our study is aiming for evaluation f the titre of anti-A and anti-B in plasma of blood grop O donors, study the effect of pooling of blood product on the level of A and B isoagglutinins in blood group O donors and screening for the safest group o donors(who have the lowest anti-A antd anti-B titre) for transfusion in urgent need of blood.

DETAILED DESCRIPTION:
the use of O blood group transfusion to patients of all groups has continued since the second world war, nevertheless the transfusion of group O plasma/ platelet concentrate to group A, B and AB recipient sometimes causes severe red cell destruction , Acute haemolysis has been reported following transfusion of non-iso group single donor platelet (PLT) concentrates and may be more common than is appreciated.

This red blood cells destruction happens based on the fact that the sera from group O people contain two separable antibodies, anti-A and anti-B .

When it comes to PLT transfusion therapy we are dealing with issues arising from the fact that PLTs contain both significant amounts of ABO antigen on their surface, as well as anti ABO isogglutinins in the donor's plasma which caused reduction the volume of incompatible plasma administrated.

From another point of view the risk of high titer units is considered low with group O, post storage, pooled PLT concentrate. However its necessary to establish a (golden standard) method for the determination of antibody titer in order to be able to differentiate accurately the high titer donors.

So, for improving the safety of group O plts we need to define a safe level of antibody titer or reduce the volume of incompatible plasma administrated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults blood group O donors

Exclusion Criteria:

* Other blood groups donors.
* Donors with history of chronic or autoimmune diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: group O donors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Decrease the risk of red cell destruction resulting from transfusion of RBCs/ platelet concentrate group O transfusion in urgent cases. | 2 years
  Using blood group typ "O" For other blood group types without causing any reaction resulting from blood transfusion .

SECONDARY OUTCOMES:
screening for the best group O donors to use for other groups urgent cases as a reserve for transfusion. | 2 years
  Using blood group typ "O" For other blood group types without causing any reaction resulting from blood transfusion .

REFERENCES:
- See also: Related Info — http://medcraveonline.com/HTIJ/HTIJ-01-00017.pdf